CLINICAL TRIAL: NCT03220087
Title: Study to Evaluate the Use of Resources and the Costs Associated With Controlled or Uncontrolled Carcinoid Syndrome in Patients With Neuroendocrine Tumours (NETs) in Spain
Brief Title: Study to Evaluate the Use of Resources and the Costs Associated With Carcinoid Syndrome (CS) in Patients With NETs in Spain
Acronym: RECOSY
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52030-367
Record Dates: First submitted 2017-06-26; First posted 2017-07-18 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A - Uncontrolled CS: Patients who have had at least one episode of uncontrolled CS, according to medical criteria, since the start of their treatment for NET.
  Interventions: Other: Data collection
- Group B - Controlled CS: Patients who have not had any episode of uncontrolled CS, according to medical criteria, in the last 12 months.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The study consists of a single visit in which socio-demographic and clinical variables will be collected from the medical record or directly from the patient. In addition, the physician will provide information on the clinical status of the disease and the patient will fill in the questionnaire.

SUMMARY:
The objective of this study is to describe the use of resources and the costs associated with controlled or uncontrolled CS in patients with NETs in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older.
* Patient with a diagnosis of NET (G1 or G2) treated with Somatostatin Analogues (SSAs) to manage their symptoms.

  1. Group A: patient who has had at least one episode of uncontrolled CS, according to medical criteria, since the start of treatment.
  2. Group B: patient who has not had any episode of uncontrolled CS, according to medical criteria, in the last 12 months.
* Patient able to read and understand the study questionnaires.
* Patient who has given written informed consent to participate in the study.

Exclusion Criteria:

* Patient participating in another clinical study when invited to participate in this study.
* Patient with another severe malignant disease.
* Patient who cannot meet the requirements established in the protocol (non-compliant or unfit to fill in the questionnaires).
* Patient with symptoms or diseases that could be confused with CS or render CS more difficult to evaluate: right cardiomyopathy or diarrhoea of any aetiology other than NET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Use of resources and costs in patients with controlled or uncontrolled CS | Day 1 (Group A retrospective data collection - 3 months before and up to 6/12 months after the last uncontrolled carcinoid episode. Group B retrospective data collection - up to 6/12 months before the date of enrolment)

SECONDARY OUTCOMES:
Clinical characteristics and therapeutic management of patients with NET and controlled or uncontrolled CS | Day 1 (Group A retrospective data collection - 3 months before and up to 6/12 months after the last uncontrolled carcinoid episode. Group B retrospective data collection - up to 6/12 months before the date of enrolment)
  A descriptive analysis of the diagnostic process; time of evolution of the disease; treatment prescribed following the diagnosis of NET and reason for choice; time elapsed from the diagnosis of NET to the first therapeutic intervention; prior and current drug treatment for NET and CS (active substance, type of treatment [rapid action vs prolonged action], dose and duration); concomitant diseases (including cardiac complications); New York Heart Association (NYHA) functional classification (I-IV); proBNP, chromogranin A and 5HIAA value; and value of the last echocardiogram, as well as any other treatments and interventions that the patient may have undergone (Yes/No, active substance and type of intervention) will be performed. The results will be compared between the two groups of patients using the paired t test for continuous variables and the Cochran-Mantel-Haenszel test or conditional logistic regression for categorical variables.
Relationship between the state of health perceived by the patient and the clinical status of the disease reported by the physician. | Day 1 (Group A retrospective data collection - 3 months before and up to 6/12 months after the last uncontrolled carcinoid episode. Group B retrospective data collection - up to 6/12 months before the date of enrolment)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (28):
- Spain (28):
  - Hospital General Univ. de Elche, Alicante
  - ICO Badalona, Badalona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital General Univ. de Ciudad Real, Ciudad Real
  - Hospital Univ. Donostia, Donostia / San Sebastian
  - Hospital Univ. de Guadalajara, Guadalajara
  - Hospital Univ. Severo Ochoa, Leganés
  - Hospital Univ. La Princesa, Madrid
  - Hospital Univ. Ramón y Cajal, Madrid
  - Hospital Clínico de San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Univ. la Paz, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital Univ. Central de Asturias, Oviedo
  - Hospital Univ. Son Espases, Palma de Mallorca
  - Hospital Montecelo, Pontevedra
  - Hospital Clín. Univ. de Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Doctor Peset, Valencia
  - Hospital la Fe de Valencia, Valencia
  - Hospital do Meixoeiro, Vigo
  - Hospital Clínico Univ. Lozano Blesa, Zaragoza
  - Hospital Univ. Miguel Servet, Zaragoza